CLINICAL TRIAL: NCT01418326
Title: Cancer Mortality Affected by the Choice of Anesthetic Drugs?
Status: Completed | Type: Observational
Sponsor: Enlund (Other)
Responsible Party: Sponsor-Investigator, Enlund, Associate professor, Uppsala University
Organization: Uppsala University (Other)
Other Study IDs: 2008350
Record Dates: First submitted 2011-05-12; First posted 2011-08-17 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer; Colo-rectal Cancer; Skin Cancer
Keywords: Cancer - breast; colo-rectal; skin
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sevoflurane: Sevoflurane exposure for radical cancer surgery
- Propofol: Propofol exposure for cancer surgery

SUMMARY:
Knowledge gap: Does the choice of anaesthetic affect outcome for cancer surgery?

Aim: To retrospectively examine possible associations (Cox Multiple Regression) between survival from breast-, colorectal-, or skin cancer and the choice of hypnotic used during surgery, ahead of a prospective randomised controlled trial.

Hypotheses: One- and five-year survival will be significantly higher after radical breast-, colorectal-, or skin cancer surgery in patients given the intravenously administered hypnotic propofol than in patients given the inhalational hypnotic sevoflurane.

Method: To merge two registers, of which one holds demographic- anaesthetic-, and surgical data from 6 303 patients operated on at the three mentioned anatomical locations at the Central Hospital in Vasteras, Sweden during a twelve year period (1998-2009). Of these minimum 4 500 operations would be due to cancer. This register is unique, in that it contains both types of anaesthesia. The other register holds survival data (date and cause of death), stored at the Regional Oncologic Center in Uppsala.

The choice of anaesthetic will be validated by controlling each patient's anaesthetic paper file, concomitantly with extraction of details from anaesthesia and surgery, such as the functional classification of each patient (according to American Association of Anesthesiologists), co-morbidity, duration of anaesthesia and surgery, amount of blood loss and possible transfusion.

Current knowledge: Different anaesthetics have opposite effects on the immune system and on the DNA. There is a well-established association between the state of the immune system and cancer growth, which in turn will influence survival. There is also an association between DNA damage and cancer development. Inhalational anaesthetics, e.g. sevoflurane, act pro-inflammatory, and they are also proven to be genotoxic. Propofol is anti-inflammatory and anti-oxidative, and it is not genotoxic.

Objective: Strengthen the hypotheses, and get statistics for a proper power calculation in advance of a multi-centre, prospective, randomised, controlled trial.

Impact: General anaesthesia is an indispensable part of radical cancer surgery. Undesired effects from anaesthesia on survival has strong relevance for the over all cancer treatment.

DETAILED DESCRIPTION:
Purpose and aims By means of record-linkage, information from two registers will be merged to retrospectively examine possible associations between survival from breast-, colorectal-, or skin cancer with the choice of hypnotic used during surgical removal of the cancer.

We hypothesize that: the one- and five-year survival rate after radical breast-, colorectal- or skin cancer surgery in general anesthesia is significantly higher in patients given the intravenously administered hypnotic propofol compared with the survival in patients exposed to the inhalational hypnotic sevoflurane.

The hypothesis is based on: 1) The knowledge about the opposite effects on the immune system from the two different anesthetics and from their different genotoxic potentials 2) The well-established associations between the state of the immune system and cancer growth, and DNA damage and cancer development, with potential influences on survival.

Survey of the field Rationale and current state of knowledge A) Immuno-modulation Converging evidence from animal studies and studies of human cell-lines indicate that different anesthetics have opposite effects on the immune system. Commonly used inhalational hypnotics are in this context pro-inflammatory, whereas the intravenously administered hypnotic agent propofol is anti-inflammatory and also anti-oxidative. A few clinical studies have indicated similar effects in patients, and a recent review has suggested that "tailoring an anesthetic plan to patient's needs will become increasingly critical, and immunology should help in this pursuit".

More specifically, previous studies have investigated the immunological effects of different anesthetics on monocytes, macrophages, natural killer cells, t-cytotoxic cells, and t-helper cells. By affecting t-helper cells anesthetics indirectly affects the production of anti-inflammatory mediators, such as interleukin-4 and -10. Anesthetics also affect the production of pro-inflammatory cytokines, such as tumor necrosis factor alpha, and interleukin-1 and -6. Moreover, the effects could be indirect by blocking or non-blocking of the surgical stress response via the hypothalamic-pituitary-adrenal axis and the sympathetic nervous system. Thus, stress hormones, such as catecholamines and cortisol, mediates inhibitory effects on immune functions. In a highly complex way, the neuroendocrine system together with both pro-inflammatory- and anti-inflammatory cytokines augments their immuno-suppressive effects. Taken together, results from previous research support that inhalational hypnotics are immuno-suppressive in mice as well as in humans.

Earlier findings also indicate other adverse effects of inhalational hypnotics that could be related to immunological processes. For example, inhalational hypnotics seem to increase the occurrence of cancer metastases. These adverse effects have not been found for propofol. In contrast, propofol seem to inhibit tumor growth and reduce the tendency to induce metastases.

The research field of immuno-modulation from anesthetics was recently reviewed by Kurosawa and Kato. They concluded, that "clinical anesthesiologists should select anesthetics and choose anesthetic methods with careful consideration of the clinical situation and the immune status of critically ill patients, in regard to long-term mortality, morbidity, and the optimal prognosis". A key note is, that "many in vitro investigations have elucidated the dose-dependent and time-dependent immunosuppressive effect of volatile (read inhalational) anesthetics on various immune cells". It was stressed in another review by Meiler, "that the perioperative process could be responsible for later adverse events", and the necessity to "understand the underlying biology and immunology should be particularly helpful in this pursuit". Thus, the choice of hypnotic may affect survival after cancer surgery. More specifically, the combined effects of surgical stress and the burden of cancer and perhaps other aggravating circumstances, such as high age and malnutrition, may play a salient role in postoperative morbidity and mortality.

B) Genotoxicity Genotoxic agents may negatively affect patient's survival after cancer surgery, as the connection between DNA damage and cancer development is well-known. The potential genotoxicity from inhalational anesthetic agents in patients and in exposed staff in operating rooms has been studied both in vitro and in vivo. A dose-response relationship for inhalational agent exposure and DNA damage has been suggested. The techniques used, the rate of sister chromatid exchange in lymphocytes and the alkaline comet assay, as indicators of genotoxicity are well validated, and they are frequently used in other contexts. Inhalational agents seem to be consistently genotoxic, whereas the less studied propofol seems not to be so.

Project description: Retrospective, follow-up cohort study.

Patients We have in an administrative system demographic-, anesthetic-, and surgical data logged by computer available for all patients exposed to anesthesia and surgery, dated from January 1, 1998 to December 31, 2009. Data includes the choice of hypnotic. All approx. 4500 patients operated on for breast-, colorectal-, or skin cancer (malignant melanoma) have been extracted from this register. Remaining demographic-, anesthetic-, and surgical data of interest will be extracted from patient's individual paper files. A data base will be constructed in the Statistical Program for Social Sciences, SPSS (Chicago, IL, USA). Accessible outcome data are stored at the Regional Oncologic Center in Uppsala.

Bias, especially potential major confounders, control of

1. The risk of selection bias is an inherent major disadvantage with a retrospective study. Here the risk is considered low due to the non-selective use of the hypnotics. Misclassification errors will be corrected on an individual level and important confounders identified at group level, c.f. down.
2. The distribution of different demographic characteristics between the two groups will be controlled for by the thorough survey of every individual patient file. Data on type and stage of the cancer, as well as different prognostic markers will also be included. Any unequal distribution of such confounders will be identified. Data on alcohol consumption will not be available.
3. Opioids also affect the immune system, and they will therefore theoretically constitute to be major confounders. This holds true for morphine, which we never use intra-operatively. Synthetic opioids, such as fentanyl, alfentanil, and remifentanil, all used by us intra-operatively, have been proven not to suppress the immune response like morphine does. On the contrary, the synthetic opioids may have positive effects in this context. We use synthetic opioids for every surgical patient at our hospital, as most other hospitals do worldwide. We have no reason to suspect an uneven administration of postoperative morphine to the two study groups, but this has also to be controlled for during data extraction.
4. Nitrous oxide, impairs the immune defense, and it also impairs DNA production by inhibition of the vitamin B12 component of methionine synthetase. Nitrous oxide will be a potential confounder for a fraction of our study population. It remains to be seen during a thorough survey of our data, if the use of nitrous oxide was evenly distributed between our two study groups?
5. Red blood cell transfusion may affect survival after cancer surgery. An immuno-suppressive effect from the allogenic material is one suggested cause. We will identify those patients having peri-operative red blood cell transfusions, control the distribution between the groups, and include them in a subgroup analysis.
6. A preceding or subsequent anesthetic given in proximity to the index procedure constitutes an important confounder and must therefore be identified. An executive decision was made defining this time span of ± 1 year from the index operation. Patients, who were anesthetized once or more than so besides the index operation within this time frame, and patients who were anesthetized from the end of the time frame to inclusion in the study will constitute separate subgroups. Accordingly, they will be analyzed separately. We assume that 10-20% of patients had another general anesthetic within the defined time interval. This assumption is based on a small pilot investigation of 100 patients in the cohort.
7. Different adjuvant cancer therapies with potent toxicity and serious side-effects will also be registered and controlled for from a confounding point of view.

Linking and matching of databases The administrative database, created as described above, will be record-linked to the regional quality registers at the Regional Oncologic Center (ROC) in Uppsala. The registers have been found to be >97% completeness compared to the Swedish Cancer Register (SCR), to which reporting is mandatory and regulated by law. The SCR holds diagnoses only and contains no clinical information. The ROC includes a quality register for breast cancer, which was started in 1992. A register for colon cancer was started in 1995, another for melanoma was started in 1996, and one for rectal cancer was created in 1997. These registers contain information on mode of detection, histopathology, stage at diagnosis, other prognostic markers and complementary treatment given. Hence, complete oncologic- and outcome data will be available for all types of cancer included in the study within the defined period of time. Data on type and stage of the cancer, as well as different prognostic markers recorded in the oncologic registers will be extracted, as well as data on recurrences of disease, vital status and date and cause of death. The unique personal identification number will be replaced by unidentified serial numbers, to ensure anonymity for each person after data securing.

Analysis The main endpoint will be a comparison of overall survival using time to event analysis. Cumulative 1- and 5-year overall survival will be assessed using the Kaplan Meier method and the estimates will be compared between patients given sevoflurane or propofol. In a next step, Cox Proportional hazard models will be calculated to assess the risk of death adjusted for potential effect modifiers and confounders. There will also be stratifications for different types of tumors, cardio-pulmonary status, ASA-class etc. Hazard ratios (HR) with 95 % confidence intervals (CI) will be presented for all models. Subgroup analyses will be undertaken for patients having more than one anesthetic within the defined time frame; a) given the same hypnotic as during the index procedure, b) given the other hypnotic at the different occasion(s); and c) for patients having one or more anesthetics outside the defined time frame.

Statistics A clinically relevant absolute difference in five-year-survival would be 5%, e.g. a difference between 85% and 80%, the latter being an average one-year-survival for the period of interest for breast cancer, which constitutes the largest group in the study. With more than 3000 patients anesthetized with sevoflurane, and more than 1000 patients anesthetized with propofol, we will have a 95% power to detect the difference with a P-value of <0.05, i.e. there will be a good margin for an unanticipated loss of data or ditto exclusions.

Ethics The project was accepted by the Regional Ethics Committee Jan 21, 2009 (2008/350). The retrospective approach will not create ethical considerations.

Significance Undesired effects from anesthesia on survival have strong relevance for the overall cancer treatment. Any suspicions of such a dramatic side-effect as potentially fatal immuno-modulation or genotoxicity must be investigated.

If the hypotheses are confirmed the results from the present study will be used for a large-scale randomized controlled trial (RCT) at multiple centers to compare the two agents, and this in turn might result in a change in practice should the results be positive. If the hypothesis is ruled out, the choice between inhalation and intravenous anesthesia will not be influenced by oncological considerations, which is important to know, although it also have to be confirmed in a RCT.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to general anesthesia for surgical removal of cancer in breast, colo-rectally, or in skin

Exclusion Criteria:

* Paper file unable to find or missing data in anesthetic file or in outcome registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients operated on for cancer in breast, colo-rectally, or in skin at a single institution from Jan 1, 1998 to Dec 31, 2009.
Sampling Method: Non-Probability Sample
Enrollment: 3284 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Survival | One year from index procedure

SECONDARY OUTCOMES:
Survival | Five years from index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mats Enlund, M.D., Ph.D., Principal Investigator — Uppsala University, Centre for Clinical Research-Vasteras; Leif Bergkvist, M.D., Ph.D., Study Director — Uppsala University, Centre for Clinnical Research-Vasteras; Mats Lambe, M.D., Ph.D., Study Chair — Uppsala University, Regional Oncologic Centre
Locations (1):
- Uppsala University, Centre for Clinical Research-Vasteras, Västerås, Sweden

REFERENCES:
- [Result] Enlund M, Berglund A, Andreasson K, Cicek C, Enlund A, Bergkvist L. The choice of anaesthetic--sevoflurane or propofol--and outcome from cancer surgery: a retrospective analysis. Ups J Med Sci. 2014 Aug;119(3):251-61. doi: 10.3109/03009734.2014.922649. Epub 2014 May 26. PMID 24857018